CLINICAL TRIAL: NCT07224386
Title: Multi-Modal Monitoring of Disease Symptoms in Myasthenia Gravis
Acronym: BioDigit MG-02
Status: Not yet recruiting | Type: Observational
Sponsor: BioSensics (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BioDigit MG-02; R44NS122672 (NIH)
Record Dates: First submitted 2025-10-29; First posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Myasthenia Gravis; Myasthenia Gravis, Generalized
Keywords: myasthenia gravis; digital health; wearable sensors
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myasthenia Gravis: All participants meeting the study inclusion criteria will be assigned to this group to complete the study activities

SUMMARY:
Evaluate the feasibility of using digital health technologies to monitor symptoms in myasthenia gravis (MG).

Study subjects will be screened and enrolled at Massachusetts General Brigham Hospital to participate in this 12 month observational study. Study subjects will be asked to wear multiple wearable sensors to monitor their physical activity and PPG during daily activities. Participants will also complete speech, video, and ePRO and eCOA digital assessments at home and during study visits.

The primary objective for this observational study is to measure the correlation of sensor-derived measures of physical activity to MG-specific ratings of MG-ADL, QMG, MGC, and Neuro-QoL Fatigue

DETAILED DESCRIPTION:
MG is a chronic autoimmune neuromuscular disease characterized by fluctuating muscle weakness that interferes with activities of daily living. Ocular, facial, swallowing, neck, limb and breathing muscles can be affected. The prevalence of MG is estimated at approximately 60,000 patients in the United States. MG symptoms are currently assessed in person through a careful history and physical exam by a neuromuscular disease expert. This is time-consuming, costly, and poses challenges in a chronic disease with fluctuating symptoms, where patients may not demonstrate any abnormality at the time of in-clinic assessment. The principal means of measuring disease severity are specific scales such as the MGC, QMG and the MG Manual Muscle Testing (MMT) scales. Although valuable, these scales are subjective and require training to administer correctly. Additionally, they provide only snapshot of a patient's disease and do not adequately reflect the spectrum of fluctuating weakness, which is a hallmark of MG. Wearable sensors and digital health technologies could enable objective, sensitive, continuous assessment of physical activity as well as motor and ocular impairments in individuals with MG.

BioSensics LLC (Newton, MA) is a medical device company specializing in wearable sensors and digital health technology for healthcare. BioSensics LLC offers a wearable sensor system and digital health solution for long-term remote monitoring of motor performance during everyday life.

The first phase of this project (NCT06277830) was conducted by Dr. Amanda Guidon at MGB, recruiting 20 patients with generalized MG over the course of 5 months to test initial feasibility of BioDigit MG.

This is an analytic observational study following participants over the course of 12 months. Subjects with documented diagnosis of MG with MGFA severity classes IIa/b, IIIa/b or IVa/b will be screened and recruited to participate in this non--interventional study.

The objective of the study is to evaluate the feasibility of using wearable sensors and digital health technologies to measure motor and speech function, as well as developing measures of ocular and facial expression to monitor the progression of the disease for people with MG. To achieve these objectives, we will conduct an observational study to investigate the correlation between outcomes as measured by the PAMSys sensor and digital health technologies with the total score and sub-scores of MG-ADL, QMG, MGC, and Fatigue Short Form of the Neuro-QOL in individuals with different MGFA severity Classes (Class IIa/b, IIIa/b or IVa/b).

ELIGIBILITY:
Inclusion Criteria:

* Autoimmune MG with or without history of thymoma, MGFA severity Class IIa/b, IIIa/b or IVa/b at the screening visit
* Diagnosed gMG through ONE of the following methods:

  * Positive acetylcholine receptor antibody (AChR Ab) test
  * Positive muscle specific kinase receptor antibody (MuSK Ab) test
  * Positive LRP4 antibody and abnormal neuromuscular transmission demonstrated by single-fiber electromyography (SFEMG) or repetitive nerve stimulation (RNS) OR has maintained a positive response to treatments such as AChE inhibitors, IVIG/PLEX, FcRn antagonists or C5 inhibitors
  * Abnormal neuromuscular transmission demonstrated by single-fiber electromyography (SFEMG) or repetitive nerve stimulation (RNS) OR has maintained a positive response to treatments such as AChE inhibitors, IVIG/PLEX, FcRn antagonists or C5 inhibitors.
* Physically and cognitively able to provide informed consent and adhere to the protocol, as determined by the investigator's judgment
* Ambulatory status defined as the ability to walk a distance of 10 meters independently, with or without the use of an assistive device
* Male or female, between the ages of 18 years old and 80 years old
* Speaks and reads English fluently

Exclusion Criteria:

* Inability to engage in activities that are essential for independent living, such as dressing, bathing, toileting, or eating independently.
* Neurological or orthopedic problems independent of myasthenia which significantly affect gait and ADLs in the investigator's judgement.
* Any significant medical, laboratory, or psychiatric condition that, in the judgment of the investigators, would potentially interfere with the ability to participate in the study.
* Residence in long-term care centers or institutions, nursing facilities, skilled nursing facilities, or recipients of hospice care, or incarceration.
* MGFA severity class I or V (MG crisis)
* Pregnant women.
* Concurrent participation in an interventional clinical trial (observational studies, biomarker studies and registries are acceptable)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with gMG with MGFA severity class IIa/b, IIIa/b or IVa/b
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in daily walking duration during activities of daily living from baseline to 12 months as measured by the PAMSys pendant | From baseline 12 months.
  Daily walking duration (hours) will be measured by the PAMSys pendant. PAMSys is a FDA-listed Class II wearable device for measuring physical activity and posture during activities of daily living.
  PAMSys will be worn for 1 week before the baseline, 3 month, 6 month, 9 month, and 12 month visits.
Change in daily number of sit to stand transitions (count) during activities of daily living from baseline to 12 months as measured by the PAMSys pendant. | From baseline to 12 months.
  Daily number of sit to stand transitions will be measured by the PAMSys pendant. PAMSys is a FDA-listed Class II wearable device for measuring physical activity and posture during activities of daily living.
  PAMSys will be worn for 1 week before the baseline, 3 month, 6 month, 9 month, and 12 month visits.

SECONDARY OUTCOMES:
Change in intelligibility when reading a standard Rainbow passage from baseline to 12 months as measured by BioDigit Speech | From baseline to 12 months.
  Speech data will be collected from participants while reading a standard Rainbow passage on a biweekly basis for 12 months. BioDigit Speech, and automatic speech analysis software, will be used to analyze the collected speech data to calculate intelligibility of speech during reading a standard Rainbow passage.
Change in Marginal Reflex Distance-1 during the upward gaze test as measured by BioDigit Video from baseline to 12 months | From baseline to 12 months.
  Video data will be collected from participants while performing a standard upward gaze test on a biweekly basis for 12 months. BioDigit Video, an automatic video analysis software, will be used to analyze the collected video data to calculate Marginal Reflex Distance-1 during the upward gaze test.
Change in total score of Myasthenia Gravis Activities of Daily Living (MG-ADL) Questionnaire from baseline to 12 months | From baseline to 12 months.
  Scores for the MG-ADL range from 0-24. A lower score represents a better outcome and a higher score is a worse outcome. Collected every two weeks.
Change in total score of the Myasthenia Garvis Composite (MGC) questionnaire from baseline to 12 months | From baseline to 12 months.
  Scores for the MGC range from 0-50. A lower score represents a better outcome and a higher score is a worse outcome. Collected every 3 months.
Change in total score of Myasthenia Gravis Quality of Life - Revised (MGQoL-15r) from baseline to 12 months | From baseline to 12 months.
  Scores for the MGQoL-15R range from 0-30. A lower score represents a better outcome and a higher score is a worse outcome. Collected every two weeks.
Change in total score of the Quantitative Myasthenia Gravis (QMG) scale from baseline to 12 months | From baseline to 12 months.
  Scores for the QMG range from 0-39. A lower score represents a better outcome and a higher score is a worse outcome. Collected every 3 months.
Change in total score of Quality of Life in Neurological Disorders - Fatigue (Neuro-QoL Fatigue) from baseline to 12 months. | From baseline to 12 months.
  Scores for the Neuro-QoL Fatigue range from 8-40. A lower score represents a better outcome and a higher score is a worse outcome. Collected every two weeks.

OTHER OUTCOMES:
Change in daily mean heart rate (beats per minute or BPM) during activities of daily living from baseline to 12 months as measured by the Samsung Galaxy watch | From baseline to 12 months.
  Heart rate will be measured during activities of daily living using the Samsung Galaxy watch.
  Samsung Galaxy watch will be worn continuously from 1 week prior to baseline until the 12 month visit.
Change in forced vital capacity during a standard spirometer breathing test from baseline to 12 months as measured by a FDA-listed spirometer | From baseline to12 months
  Forced vital capacity (FVC) will be measured directly by the spirometer during a standard breathing assessment. The FVC will be measured in Litres. FVC will be collected biweekly from baseline to 12 months
Change in articulatory rate when reading a standard Rainbow passage from baseline to 12 months as measured by BioDigit Speech | From baseline to 12 months
  Speech data will be collected from participants while reading a standard Rainbow passage on a biweekly basis for 12 months. BioDigit Speech, and automatic speech analysis software, will be used to analyze the collected speech data to calculate articulatory rate during reading a standard Rainbow passage.
Change in eye aspect ratio during the upward gaze test as measured by BioDigit Video from baseline to 12 months | From baseline to 12 months.
  Video data will be collected from participants while performing a standard upward gaze test on a biweekly basis for 12 months. BioDigit Video, an automatic video analysis software, will be used to analyze the collected video data to calculate eye aspect ratio during the upward gaze test.
Change in daily mean heart rate variability during activities of daily living from baseline to 12 months as measured by the Samsung Galaxy watch | From baseline to 12 months.
  Heart rate variability will be measured during activities of daily living using the Samsung Galaxy watch.
  Samsung Galaxy watch will be worn continuously from 1 week prior to baseline until the 12 month visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Neuromuscular Diagnostic Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Mishra RK, Potter IY, Enriquez A, Stafstrom CL, Sheitman Z, Lindsay A, Barchard G, Nunes AS, Duda PW, Vaziri A, Guidon AC. Development and Feasibility Assessment of a Multimodal Digital Health Technology for Remote Monitoring of Symptoms in Myasthenia Gravis. Digit Biomark. 2025 Oct 23;9(1):193-202. doi: 10.1159/000549122. eCollection 2025 Jan-Dec. PMID 41322084